CLINICAL TRIAL: NCT00274859
Title: Multicenter Phase II Study Evaluating Gemcitabine and Oxaliplatin in the Treatment of Patients Suffering From Metastatic Breast Cancer Who Are Not Candidates For Treatment With Antracyclines and Taxanes
Brief Title: Gemcitabine and Oxaliplatin in Treating Patients With Metastatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454320; GERCOR-SEGEMOX-S04-1; LILLY-GERCOR-SEGEMOX-S04-1; SANOFI-GERCOR-SEGEMOX-S04-1; EU-20571
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with oxaliplatin works in treating patients with metastatic cancer who cannot receive anthracycline or taxane therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with metastatic cancer not amenable to anthracycline or taxane therapy treated with gemcitabine hydrochloride and oxaliplatin.

Secondary

* Determine the clinical benefit and tolerability of this regimen in these patients.
* Determine the progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive gemcitabine hydrochloride IV over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer

  * Metastatic disease
* Measurable metastatic disease ≥ 1 cm by spiral CT scan and/or cutaneous lesion ≥ 2 cm
* Not a candidate for anthracycline or taxane chemotherapy
* No brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Alkaline phosphatase < 5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Creatinine < 1.5 times ULN OR creatinine clearance > 30 mL/min
* SGOT and SGPT < 3 times ULN (5 times ULN if liver metastases present)
* No pre-existing neuropathy
* Not pregnant or nursing
* No uncontrolled hypercalcemia
* No familial, social, geographical, or psychological condition that would preclude study treatment
* No other malignancy that is not considered cured

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease, including anthracyclines or taxanes
* Prior hormonal therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2005-08

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Clinical benefit
Tolerability
Progression-free
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gligorov, MD, Study Chair — Hopital Tenon
Locations (14):
- France (14):
  - C.H.G. Beauvais, Beauvais
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - Centre Jean Perrin, Clermont-Ferrand
  - Intercommunal Hospital, Montfermeil
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Polyclinique De Courlancy, Reims
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - C.H. Senlis, Senlis
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier Intercommunal Toulon - La Seyne Sur Mer, Toulon
  - Institut Gustave Roussy, Villejuif